CLINICAL TRIAL: NCT05066100
Title: Prenatal Diagnosis and Treatment of Flat, Inverted and Retracted Nipples to Improve Postpartum Breastfeeding Rates
Brief Title: Prenatal Diagnosis and Treatment of Flat, Inverted and Retracted Nipples
Acronym: FIRN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not started due to administrative considerations.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Miriam (Miri) E. Levi, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-006665
Record Dates: First submitted 2021-09-06; First posted 2021-10-04 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Inverted Nipple; Retracted Nipple
Keywords: Pregnancy; Lactation; Postpartum; Flat Nipples; Inverted Nipples; Retracted Nipples
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women with FIRN (Experimental): Women desiring to breastfeed and identified during their pregnancy as having flat, inverted or retracted nipples
  Interventions: Other: Prenatal Use of Supple Cups

INTERVENTIONS:
Other: Prenatal Use of Supple Cups — For pregnant women identified with FIRN and providing consent to participate in this study, Supple Cup usage will be initiated at 32 weeks gestation to begin to elongate the nipples in preparation for breastfeeding.

SUMMARY:
The objectives of this study are to determine the population occurrence rate of flat, inverted, or retracted nipples (FIRN) in pregnant women in our obstetrical practice through prenatal evaluation at the NOB visit and re-evaluation at the 28th-30th week of gestation, to determine the benefit of using Supple Cups as treatment for FIRN for 6-8 weeks in the third trimester to evert the nipples prior to delivery, and to evaluate the effect of prenatal diagnosis and treatment of FIRN on establishment of latch and breastfeeding rates in the postpartum period.

DETAILED DESCRIPTION:
It is well established that breastfeeding is the most clinically optimal method of feeding for infants through the first year of life, however exclusive breastfeeding rates in the United States remain low. Many women have difficulty establishing breastfeeding in the first few weeks after birth which leads to the use of formula supplementation. For approximately 10% of women this difficulty is caused by flat, inverted or retracted nipples (FIRN) which make it very difficult to latch when attempting to breastfeed. Many women are not diagnosed with FIRN until after the baby is born.

Supple Cups are promising as a prenatal and postnatal intervention to elongate nipples in cases of FIRN, allowing women with these biological variations to successfully breastfeed. If women are diagnosed in the early prenatal period with FIRN, Supple Cup use can be initiated to elongate and prepare the nipples for breastfeeding postpartum. Pre-natal diagnosis of FIRN is critical to enable breastfeeding immediately postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* Pregnant at time of enrollment
* Plan to breastfeed their infant following birth
* Plan delivery at Mayo Clinic Hospital
* One or more flat, inverted or retracted nipple diagnosed by a healthcare professional

Exclusion Criteria:

* History of breast surgery or nipple piercings
* History of significant low milk supply requiring discontinuation of breastfeeding prior to six weeks postpartum
* History of preterm labor and/or birth
* History of high-risk medical condition that increases patient risk for preterm labor and/or birth
* History of Raynaud's syndrome and/or hypersensitivity to palpation of breasts
* Current multiple gestation pregnancy
* Active rash, infection, or lesions on the nipple at time of initiation of Supple Cups

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Percent of women with change in nipple elongation following use of Supple Cups in the prenatal period | At completion of 6 weeks of Supple Cups use during the prenatal period
  Visual assessment and documented description of change in elongation of nipple after using Supple Cups prior to birth

SECONDARY OUTCOMES:
Percent of women with established breastfeeding with adequate infant latch | One week postpartum
  Visual assessment and documentation of a consistent infant latch during breastfeeding for the women who utilized Supple Cups in the prenatal period.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam E Levi, CNM, MBA, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota, United States